CLINICAL TRIAL: NCT00692133
Title: Spanish Validation of Tool Questionnaire to Assess Patients´Perception About Antipsychotic Treatment
Acronym: TOOL
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Teresa Díez, AstraZeneca Pharmaceuticals
Other Study IDs: NIS-NES-DUM-2007/2
Record Dates: First submitted 2008-06-05; First posted 2008-06-06 (Estimated); Last update posted 2010-12-10 (Estimated); Status verified 2010-12

CONDITIONS: Schizophrenia; Bipolar Disorder
Keywords: schizophrenia; bipolar disorder; antipsychotic treatment; patients´preferences
MeSH Terms: conditions — Schizophrenia; Bipolar Disorder

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Non-interventional, prospective study to validate Spanish version of TOOL questionnaire in patients with schizophrenia and bipolar disorder under antipsychotic treatment

ELIGIBILITY:
Inclusion Criteria:

* Schizophrenia and bipolar disorder (DSM-IV criteria)
* Stabilized out-patients
* Treated with the same oral antipsychotic at least in the last month

Exclusion Criteria:

* Participation in another clinical trial within 6 months prior to enrolment into this study
* Administration of a depot antipsychotic medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient aged 18-year old or older who has been diagnosed as schizophrenia or bipolar disorder
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2008-03; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
TOOL questionnaire | 15 days
PANSS & Young Mania Scale | 15 days

SECONDARY OUTCOMES:
Montgomery Asberg Depression Scale | 15 days
Euroqol 5D & SF-36D | performed only at baseline visit
UKU modified scale | performed only at baseline visit

CONTACTS AND LOCATIONS:
Overall Officials: Angel L Montejo, Study Chair — University of Salamanca
Locations (32):
- Spain (32):
  - Research Site, Vitoria-Gasteiz, Alava
  - Research Site, Palma, Balearic Islands
  - Research Site, Gavà, Barcelona
  - Research Site, Burgos, Burgos
  - Research Site, Puerto Real, Cadiz
  - Research Site, Santander, Cantabria
  - Research Site, Castellon, Castellon
  - Research Site, Ceuta, Ceuta
  - Research Site, A Coruña, Coruna
  - Research Site, Atarfe, Granada
  - Research Site, Granada, Granada
  - Research Site, Arrasate / Mondragón, Guipuzcoa
  - Research Site, Donostia / San Sebastian, Guipuzcoa
  - Research Site, Linares, Jaen
  - Research Site, León, Leon
  - Research Site, Alcobendas, Madrid
  - Research Site, Madrid, Madrid
  - Research Site, Parla, Madrid
  - Research Site, Estepona, Malaga
  - Research Site, Málaga, Malaga
  - Research Site, Murcia, Murcia
  - Research Site, Elizondo, Navarre
  - Research Site, Pamplona, Navarre
  - Research Site, Tudela, Navarre
  - Research Site, Pontevedra, Pontevedra
  - Research Site, Oviedo, Principality of Asturias
  - Research Site, Salamanca, Salamanca
  - Research Site, Tarragona, Tarragona
  - Research Site, Alzira, Valencia
  - Research Site, Sagunto, Valencia
  - Research Site, Galdako, Vizcaya
  - Research Site, Zamudio, Vizcaya